CLINICAL TRIAL: NCT00020332
Title: A Phase I/II Trial of Docetaxel Followed by Infusional Flavopiridol Over 72 Hours in Patients With Previously Treated Locally Advanced or Metastatic Breast Cancer
Brief Title: Docetaxel and Flavopiridol in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068292; NCI-00-C-0212; NCI-952; NCT00006277 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2002-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — alvocidib; Docetaxel

INTERVENTIONS:
Drug: alvocidib
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy in treating patients who have locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of docetaxel and flavopiridol in patients with previously treated locally advanced or metastatic breast cancer.
* Determine the dose-limiting toxicity, toxicity profile, and pharmacokinetics of this regimen in these patients.
* Determine the activity of this regimen in these patients.
* Determine the objective response rate in patients treated with this regimen.
* Determine immune dysfunction produced by this regimen as measured by lymphocyte subpopulations, including T-cell activation/memory subsets and natural killer cell/lymphokine-activated killer cell functional subsets in these patients.
* Determine the ability of positron emission tomography scanning to predict response in patients treated with this regimen.
* Determine the response duration, time to treatment failure, and overall survival of patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.
* Determine whether this regimen is associated with the development of a prothrombotic state in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive docetaxel IV over 1 hour on day 1 followed by flavopiridol IV over 1 hour or IV continuously on days 2-4. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Sequential dose escalation of docetaxel is preceded or followed by sequential dose escalation of flavopiridol. Cohorts of 3-6 patients receive escalating doses of docetaxel preceded or followed by escalating doses of flavopiridol until the maximum tolerated dose (MTD) of the combination is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 22 additional patients are accrued to receive flavopiridol and docetaxel at the recommended phase II dose.

Quality of life is assessed at baseline, every 3 courses during study, and then at completion of study.

PROJECTED ACCRUAL: A total of 49 patients (27 for phase I and 22 for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV adenocarcinoma of the breast
* Phase I:

  * Evaluable disease allowed
* Phase II:

  * At least 1 site of measurable disease
* No bone metastasis as only site of disease
* No carcinomatous meningitis or brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No active coagulopathy requiring therapeutic anticoagulation

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than 1.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No Gilbert's disease

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* Left ventricular ejection fraction at least 50% without clinical signs or symptoms of heart failure
* No uncontrolled hypertension (sustained systolic blood pressure (BP) greater than 180 mm Hg or diastolic BP greater than 100 mm Hg)
* No uncontrolled cardiac arrhythmia
* No myocardial infarction within the past year
* No significant ischemia or valvular heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical or psychiatric condition that would increase risk
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanomatous skin cancer
* No grade 2 or greater peripheral neuropathy
* No diabetes mellitus with a fasting blood sugar greater than 200 mg/dL
* No active unresolved infection
* No serious concurrent medical illness
* No history of hypersensitivity reaction to products containing polysorbate 80 (Tween 80)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior flavopiridol
* Prior adjuvant chemotherapy for advanced disease allowed if within 6 months of diagnosis of metastatic disease
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosourea or 8 weeks for UCN-01) and recovered
* Phase I:

  * Any number of prior chemotherapy regimens for metastatic carcinoma of the breast allowed
* Phase II:

  * No more than 2 prior chemotherapy regimens for metastatic carcinoma of the breast

Endocrine therapy:

* Prior hormonal therapy in the metastatic or adjuvant setting allowed
* At least 2 weeks since prior hormonal therapy and no evidence of disease improvement by radiography after therapy
* Concurrent corticosteroids allowed if for study premedication or hypersensitivity reactions/adverse events

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent antineoplastic therapies
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette R. Tan, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States